CLINICAL TRIAL: NCT06193382
Title: Parent-Child Interaction Therapy (PCIT) for Children With Traumatic Brain Injury (TBI): A Stepped-Care Model
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Miami (Other)
Responsible Party: Principal Investigator, Dainelys Garcia, Associate Professor of Clinical Pediatrics, University of Miami
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 20230405
Record Dates: First submitted 2023-12-21; First posted 2024-01-05 (Actual); Last update posted 2025-08-26 (Actual); Status verified 2025-08

CONDITIONS: Traumatic Brain Injury; Disruptive Behavior
MeSH Terms: conditions — Brain Injuries, Traumatic; Problem Behavior

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- PCIT Group (Experimental): Participants in this group will receive the PCIT intervention for up to 5 weeks.
  Interventions: Behavioral: PCIT

INTERVENTIONS:
Behavioral: PCIT — Participants will receive the adapted Pocket PCIT Online via a web-based learning platform for up to 5 weeks. Participants will engage in this intervention weekly for about 1 hour per week. During engaging with the adapted Pocket PCIT Online version of PCIT, caregivers will learn positive parenting skills to increase the warmth of the parent-child relationship as well as strategies to effectively set limits. Participants will also participate in 15-minute check-in phone calls with a therapist each week throughout the course of treatment.
  Other Names: Step-Up PCIT; Pocket PCIT

SUMMARY:
The purpose of this study is to understand how a stepped-care model of Parent-Child Interaction Therapy (Step-Up PCIT) addresses child behavioral problems among children between the ages of 2 and 7 with a traumatic brain injury (TBI).

ELIGIBILITY:
Child Inclusion Criteria:

* Child is between the ages of 2 and 7
* Child has a mild to moderate TBI

Primary Caregiver Inclusion Criteria:

* Primary caregiver is 18 years or older
* Primary caregiver speaks and reads in either English or Spanish

Child Exclusion Criteria:

- Children with major sensory impairments (e.g., deafness, blindness)

Primary Caregiver Exclusion Criteria:

- Primary caregiver with major sensory impairments (e.g., deafness, blindness)

Min Age: 2 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2025-11-01 (Estimated); Primary Completion 2026-11-01 (Estimated); Study Completion 2026-12-30 (Estimated)

PRIMARY OUTCOMES:
Change in child behavior problem frequency and severity as measured by the Eyberg Child Behavior Inventory (ECBI) intensity scale | Baseline and week 5
  The ECBI questionnaire will be used to evaluate the number of behavioral problems and the frequency of their occurrence before and after the intervention program. ECBI provides a list of 36 problem behaviors commonly reported by parents. The inventory assesses behavior on two dimensions: 1) the frequency of the behavior; 2) whether parents consider it a problem. The frequency ratings range from 1 (never) to 7 (always), and are summed up to arrive at an overall problem behavior Intensity Score, ranging from 36 to 252. Higher score means more behavioral problems.
Change in caregiver-perceived child behavior problems as measured by the Eyberg Child Behavior Inventory (ECBI) problem scale | Baseline and week 5
  The ECBI questionnaire will be used to evaluate the number of behavioral problems and the frequency of their occurrence before and after the intervention program. ECBI provides a list of 36 problem behaviors commonly reported by parents. The inventory assesses behavior on two dimensions: 1) the frequency of the behavior; 2) whether parents consider it a problem. The frequency ratings range from 1 (never) to 7 (always), and are summed up to arrive at an overall problem behavior Intensity Score, ranging from 36 to 252. Higher score means more behavioral problems.
Change in parent stress as measured by the Parenting Stress Index Fourth Edition Short Form (PSI-SF) total score | Baseline and week 5
  PSI-4-SF assesses the parents stress level. PSI-4-SF contains 36 items: 12 items for Parental Stress (PS), 12 items for Parent-Child Dysfunctional Interaction (P-CDI), and 12 items for Difficult Child (DC).The normal range for scores is within the 16th to 84th percentiles.Scores in the 85th to 89th percentile are considered high, and scores in the 90th percentile or higher are considered clinically significant.
Change in parent stress as measured by the Parenting Stress Index Fourth Edition Short Form (PSI-SF) Parent Stress (PS) score | Baseline and week 5
  PSI-4-SF assesses the parents stress level.PSI-4-SF contains 36 items: 12 items for Parental Stress (PS) , 12 items for Parent-Child Dysfunctional Interaction (P-CDI), and 12 items for Difficult Child (DC).The normal range for scores is within the 16th to 84th percentiles.Scores in the 85th to 89th percentile are considered high, and scores in the 90th percentile or higher are considered clinically significant.
Change in parent-child dysfunctional interaction as measured by the Parenting Stress Index Fourth Edition Short Form (PSI-SF) Parent-Child Dysfunctional Interaction (P-CDI) score | Baseline and week 5
  PSI-4-SF assesses the parents stress level.PSI-4-SF contains 36 items: 12 items for Parental Stress (PS) , 12 items for Parent-Child Dysfunctional Interaction (P-CDI), and 12 items for Difficult Child (DC).The normal range for scores is within the 16th to 84th percentiles.Scores in the 85th to 89th percentile are considered high, and scores in the 90th percentile or higher are considered clinically significant.
Change in how the caregiver perceptions about how it is to care for the child as measured by the Parenting Stress Index Fourth Edition Short Form (PSI-SF) Difficult Child (DC) score | Baseline and week 5
  PSI-4-SF assesses the parents stress level.PSI-4-SF contains 36 items: 12 items for Parental Stress (PS) , 12 items for Parent-Child dysfunctional Interaction (P-CDI), and 12 items for Difficult Child (DC).The normal range for scores is within the 16th to 84th percentiles.Scores in the 85th to 89th percentile are considered high,and scores in the 90th percentile or higher are considered clinically significant.
Change in parenting skills as measured by the Dyadic Parent-Child Interaction Coding System-Fourth Edition (DPIC-IV) | Baseline and week 5
  The Dyadic Parent-Child Interaction Coding System-4th Ed is a structured behavioral observation coding system assessing caregiver-child interactions. Observed parenting behaviors will be coded during a 5-min parent-child play session with a tablet with educational apps and combined into two categories of positive (praises, behavior descriptions, and reflections) and negative (questions, commands, and negative talk) verbalizations, reflecting behaviors caregivers are taught to use and avoid in PCIT. The higher the score the higher quality the parenting behavior.
Treatment satisfaction as measured by the Therapist Attitude Inventory (TAI) | Up to 5 weeks
  TAI is a valid index of consumer satisfaction for participants in behavioral parent training (BPT). Items are rated on a scale from one (indicating treatment dissatisfaction or lack of improvement) to five (indicating satisfaction with treatment and improvement). Parents will complete this form after the last session of the BPT program. BPT consists of 11 items that are scored on a 5-point Likert scale. The total score range is 11-55; the higher the score, the greater the satisfaction
Number of modules completed by the caregiver | Up to 5 weeks
  Number of modules completed by the caregiver
Number of week homework was completed by the caregiver | Up to 5 weeks
  Number of week homework was completed by the caregiver
Acceptability of Intervention Measure (AIM) | Up to 5 weeks
  The Likert scale has 4 items. The scores will be summed to provide a total score. Scores range from completely disagree to completely agree.
Intervention Appropriateness Measure (IAM) | Up to 5 weeks
  The Likert scale has 4 items. The scores will be summed to provide a total score. Scores range from completely disagree to completely agree.
Feasibility of Intervention Measure (FIM) | Up to 5 weeks
  The Likert scale has 4 items. The scores will be summed to provide a total score. Scores range from completely disagree to completely agree.

SECONDARY OUTCOMES:
Change in family functioning as measure by the General Functioning (GF) Scale | Baseline and week 5
  The general functioning scale is made up of 12 items with six items that reflect healthy family functioning and the other six items reflecting unhealthy functioning. Scoring is on a 4-point scale (from 1 for strongly agree to 4 for strongly disagree) with the scoring for the negatively worded items reversed.
Change in child's functioning as measured by the Strengths and Difficulties Questionnaire (SDQ) | Baseline and week 5
  SDQ is a brief emotional and behavioral screening questionnaire for children and young people. Scores range from minimal value (not true) to maximum value (certainly true).The scores will be summed to provide a total score.
Change in child's emotional symptoms as measured by the Strengths and Difficulties Questionnaire (SDQ) emotional symptoms scale | Baseline and week 5
  SDQ is a brief emotional and behavioral screening questionnaire for children and young people. Scores range from minimal value (not true) to maximum value (certainly true).The scores will be summed to provide a total score.
Change in child's conduct problems as measured by the Strengths and Difficulties Questionnaire (SDQ) conduct problems scale | Baseline and week 5
  SDQ is a brief emotional and behavioral screening questionnaire for children and young people. Scores range from minimal value (not true) to maximum value (certainly true).The scores will be summed to provide a total score.
Change in child's hyperactivity/inattention as measured by the Strengths and Difficulties Questionnaire (SDQ) hyperactivity/inattention scale | Baseline and week 5
  SDQ is a brief emotional and behavioral screening questionnaire for children and young people. Scores range from minimal value (not true) to maximum value (certainly true).The scores will be summed to provide a total score.
Change in child's peer relationship problems as measured by the Strengths and Difficulties Questionnaire (SDQ) peer relationship problems scale | Baseline and week 5
  SDQ is a brief emotional and behavioral screening questionnaire for children and young people. Scores range from minimal value (not true) to maximum value (certainly true).The scores will be summed to provide a total score.
Change in child's prosocial behaviors as measured by the Strengths and Difficulties Questionnaire (SDQ) prosocial behavior scale | Baseline and week 5
  SDQ is a brief emotional and behavioral screening questionnaire for children and young people. Scores range from minimal value (not true) to maximum value (certainly true).The scores will be summed to provide a total score.

CONTACTS AND LOCATIONS:
Overall Officials: Dainelys Garcia, PhD, Principal Investigator — University of Miami; Jason F Jent, PhD, Principal Investigator — University of Miami; Jennifer Coto, PhD, Principal Investigator — University of Miami
Locations (1):
- University of Miami, Miami, Florida, United States

IPD SHARING:
Plan to Share IPD: No